CLINICAL TRIAL: NCT05425836
Title: A Randomized Controlled Trial to Compare High Flow Nasal Cannula With Standard Nasal Cannula to Prevent Desaturation in Subjects Undergoing Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS-TBNA)
Brief Title: HFNC Versus SOT During EBUS
Acronym: NOT-EBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT/IEC/2021/SPL-1049
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Endobronchial Ultrasound

STUDY DESIGN:
Intervention Model Description: Two arm parallel group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen supplementation in the conventional arm (Active Comparator): will be delivered by nasal cannula. At 5 minutes prior to sedation the flow rate would be kept a 5 L/minute.; The flow will be increased to 6-8 L/minute to maintain SPO2 ≥92% during the procedure, up to a maximum of 15 L/minute, depending on the patient tolerance.
  Interventions: Device: Standard oxygen therapy
- Oxygen supplementation in HFNC arm (Experimental): HFNC (OptiFlowTM; Fisher & Paykel, Auckland, New Zealand) will be started 5 minutes before the sedation at a flow rate of 30 Litres/minute and at a fraction of inspired oxygen (FiO2) of 0.30, which will be titrated by increments of 10 liters/minute depending on oxygen demand to keep SPO2 ≥92% during the procedure. The flow rate will be maintained between 30- and 70-liters minute, depending on the patient tolerance.
  Interventions: Device: HFNC

INTERVENTIONS:
Device: Standard oxygen therapy — nasal cannula
  Arms: Oxygen supplementation in the conventional arm
Device: HFNC — High flow nasal cannula
  Arms: Oxygen supplementation in HFNC arm

SUMMARY:
Endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration (TBNA) is a routine procedure that is performed to sample mediastinal lymph nodes. At author's center the EBUS-TBNA procedure is performed under conscious sedation using midazolam. During the EBUS procedure, oxygen supplementation can either be provided using low flow or high flow through a nasal cannula.

The investigators hypothesize that the use of high flow nasal cannula (HFNC) for oxygen supplementation during EBUS would be associated with lesser incidence of clinically significant hypoxemia (SpO2 ≤90%) when compared to conventional nasal cannula. In this study, the authors plan to assess the efficacy of HFNC in reducing the incidence of hypoxemic events in subjects undergoing EBUS under conscious sedation.

DETAILED DESCRIPTION:
Endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration (TBNA) is a routine procedure that is performed to sample mediastinal lymph nodes. The procedure is performed either under conscious sedation or using general anaesthesia. At author's center the EBUS-TBNA procedure is performed under conscious sedation using midazolam.During the EBUS procedure, oxygen supplementation is provided to prevent desaturation events. However, despite oxygen supplementation previous studies have reported fall in pulse oximetric saturation (SpO2) below 90%.

The high-flow nasal cannula (HFNC) is a novel device for providing oxygen supplementation. It delivers a flow of 10-70 litres/min of humidified, warmed 100% oxygen through a nasal cannula. The device has been used extensively in intensive care setting in adults with hypoxemic respiratory failure. In a study conducted on patients undergoing EBUS-TBNA, the use of HFNC led to a significant reduction in the number of subjects experiencing clinically significant hypoxemia (SpO2 ≤90%) compared to conventional oxygen supplementation. However, the study conclusions were limited by a small sample size. Another study demonstrated lesser episodes of hypoxemia with HFNC compared to the conventional oxygen supplementation. This study also had a small sample size (n=40). The investigators that the use of HFNC for oxygen supplementation during EBUS would be associated with lesser incidence of clinically significant hypoxemia (SpO2 ≤90%) when compared to conventional nasal cannula. In this study, the authors intend to assess the efficacy of HFNC in reducing the incidence of hypoxemic events in subjects undergoing EBUS under conscious sedation.

ELIGIBILITY:
Inclusion Criteria:

1. All adult (aged between 18 and 80 years) subjects undergoing the EBUS-TBNA procedure and pulse oximetric SPO2 ≥95% at room air will be eligible for this study

Exclusion Criteria:

1. oxygen supplementation required to achieve SPO2 >95%;
2. subjects who have altered mentation;
3. pregnancy
4. failure to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
proportion of subjects experiencing oxygen desaturation events | 1 hour (during the EBUS procedure)
  oxygen desaturation events (defined SpO2 <90% for at least 10 seconds) during the EBUS-TBNA procedure

SECONDARY OUTCOMES:
SPO2 after pre-oxygenation | 1 hour (during the EBUS procedure)
  Pre-oxygenation for 5 minutes before sedation
number of desaturation events (SPO2 <90% for at least 10 seconds) during the procedure | 1 hour (during the EBUS procedure)
  Desaturation events will defined as SPO2 <90% for at least 10 seconds
nadir SPO2 level during the procedure | 1 hour (during the EBUS procedure)
  lowest oxygen saturation
patient comfort and bronchoscopist satisfaction score | 1 hour (during the EBUS procedure)
  assessed on a visual analogue scale (VAS); VAS will be measured on a scale of 0 to 100 mm, 0 being very comfortable or satisfied and 100 being extremely uncomfortable or unsatisfied
number of participants experiencing complications in each group | 1 hour (during the EBUS procedure)
  cardiac arrhythmia, hypotension, escalation of the level of care (hospitalization, airway intubation need for non-invasive or invasive mechanical ventilation), altered mentation, respiratory failure or cardiac arrest

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Bronchoscopy suite, PGIMER, Chandigarh
  - Bronchoscopy suite, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on request to the corresponding author